CLINICAL TRIAL: NCT04358315
Title: Consumer Assessment of Tobacco Flavor and Odor
Status: Terminated | Type: Observational
Why Stopped: PI request
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: I 80518; NCI-2019-06320 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 80518 (Other: Roswell Park Cancer Institute); U54CA228110 (NIH)
Record Dates: First submitted 2020-04-13; First posted 2020-04-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Current Vaper; Healthy Subject
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (smell or puff e-liquids): All panel participants smell and user panelists puff flavored e-liquids and answer questions about the products.
  Interventions: Behavioral: Behavioral Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Smell or puff e-liquids
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies consumer assessments of tobacco flavor and odor. This study will compare the ability of expert and consumer panels to identify and characterize flavors, determine threshold detection levels for individual and mixed flavors, and identify the dominant flavor of mixtures.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Develop consumer (untrained) sensory panels to identify and assess characterizing flavors in electronic (e)-liquids.

OUTLINE:

Non-user panelists smell and user panelists puff flavored e-liquids and answer questions about the products.

ELIGIBILITY:
Inclusion Criteria:

* CONSUMER USER: Current daily vapers of products containing nicotine
* CONSUMER USER: No concurrent use of other tobacco products
* CONSUMER USER: General good health
* CONSUMER USER: No allergies
* CONSUMER USER: No self-reported taste or smell deficits
* CONSUMER USER: Not pregnant or lactating
* CONSUMER USER: No medications known to interfere with taste/smell
* CONSUMER USER: Passing scores on the Brief Smell Identification Test (B-SIT), phenylthiocarbamine (PTC) and 6-n-propylthiouracil (PROP) smell and taste tests
* CONSUMER USER: No positive diagnosis of COVID-19 within 30 days
* CONSUMER NONUSER: No use of tobacco or nicotine products in the last year
* CONSUMER NONUSER: General good health
* CONSUMER NONUSER: No allergies
* CONSUMER NONUSER: No self-reported taste or smell deficits
* CONSUMER NONUSER: Not pregnant or lactating
* CONSUMER NONUSER: No medications known to interfere with taste/smell
* CONSUMER NONUSER: Passing scores on the Brief Smell Identification Test (B-SIT), phenylthiocarbamine (PTC) and 6-n-propylthiouracil (PROP) smell and taste tests
* CONSUMER NONUSER: No positive diagnosis of COVID-19 within 30 days

Exclusion Criteria:

* CONSUMER USER: Outside age range
* CONSUMER USER: Not current daily vapers
* CONSUMER USER: Concurrent use of other tobacco products
* CONSUMER USER: Fair or poor general health
* CONSUMER USER: Allergies
* CONSUMER USER: Self-reported taste or smell deficits
* CONSUMER USER: Pregnant or lactating
* CONSUMER USER: Medications known to interfere with taste/smell
* CONSUMER USER: Failing scores on the Brief Smell Identification Test (B-SIT), phenylthiocarbamine (PTC) and 6-n-propylthiouracil (PROP) smell and taste tests
* CONSUMER USER: Positive diagnosis of COVID-19 within 30 days
* CONSUMER NONUSER: Outside age range
* CONSUMER NONUSER: Use of tobacco or nicotine products in the last year
* CONSUMER NONUSER: Fair or poor general health
* CONSUMER NONUSER: Allergies
* CONSUMER NONUSER: Self-reported taste or smell deficits
* CONSUMER NONUSER: Pregnant or lactating
* CONSUMER NONUSER: Medications known to interfere with taste/smell
* CONSUMER NONUSER: Failing scores on the Brief Smell Identification Test (B-SIT), phenylthiocarbamine (PTC) and 6-n-propylthiouracil (PROP) smell and taste tests
* CONSUMER NONUSER: Positive diagnosis of COVID-19 within 30 days

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Current daily vapers and nonusers in the greater Buffalo and Rochester areas
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Flavor identification and evaluation | Up to 12 months
  Subjects will be asked to identify various concentrations of flavored e-liquids
Specific flavor detection thresholds | Up to 12 months
  Subjects will rate intensity of odors of e liquids
Flavor combination thresholds | Up to 12 months
  Subjects will rate a combination of two e-liquids combined

CONTACTS AND LOCATIONS:
Overall Officials: Richard J O'Connor, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States